CLINICAL TRIAL: NCT05850663
Title: Quality of Life Assessment of Hypofractionated Radiotherapy in Recurrent Head and Neck Cancer: CPC-CT Pilot
Brief Title: Quality of Life Assessment of Radiotherapy in Recurrent Head and Neck Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to lack of accrual.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Quadshot mHealth
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Gynecologic Cancer; Cervical Cancer; Endometrial Cancer
Keywords: Radiation Therapy; Mobile Health; QUADSHOT; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ecological Momentary Assessments (EMAs) (Other): Patients will receive one EMA (Ecologic Momentary Assessment) per day for approximately 75 days, through the provided smart phone application.
  Interventions: Other: Ecologic Momentary Assessment (EMA)

INTERVENTIONS:
Other: Ecologic Momentary Assessment (EMA) — EMA enables measurement of phenomena in real-time, natural settings.
  EMA data will be used to identify moments of high distress, assess cancer treatment side effects, and assess barriers to care.
  The EMA methodology used in this study will ask about current emotional, physical, behavioral, and social states.
  The EMAs will consist of time-based sampling (i.e. a daily dairy), which will be prompted and initiated by the phone.

SUMMARY:
The purpose of this study is to examine the uses of a mobile health-based assessment and symptom monitoring platform.

DETAILED DESCRIPTION:
This study will involve patients who have been diagnosed with head and neck or gynecologic cancers and are receiving radiation treatments via the QUAD shot regimen. It is a single arm pilot trial designed to provide information on the ease of use, feasibility, and perceived usefulness of a smartphone application to monitor symptoms and quality of life during cancer treatment, as well as assess barriers to care and perceptions of the smartphone app.

Patients will download the study app onto their personal smartphone, if the phone is compatible with the app, or a study smartphone will be loaned to them. The smartphone app will first ask patients to complete the 15-25 minute baseline survey, followed by one daily brief survey that ask about symptoms, quality of life, and barriers for 75 days. At the end of this period, the smartphone app will prompt the patient to complete a final survey, followed by a brief in-person or telephone interview to assess opinions about the app. Patients' symptoms, treatment effects, medication adherence, pain, quality of life, and general barriers to care will be assessed with questionnaires to measure the impacts of the mobile health-based assessment platform. Results from this study will be for research only and will not impact treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Written informed consent and any locally-required authorization obtained from the patients prior to performing any protocol-related procedures, including screening evaluations
* Pathologically (histologically or cytologically) proven diagnosis of cancer of the head and neck (nasopharynx, oral cavity, oropharynx, hypopharynx, larynx, or unknown primary) or Gynecologic cancers (cervical and endometrial)
* Locally recurrent or metastatic HNC or Gyn cancer not deemed amenable to curative-intent salvage therapy, in whom at least six months have passed since their prior RT, if received
* Must have evaluable lesion per RECIST v1.1
* Patients agree to provide their smoking history prior to registration
* ECOG performance status of 0-2

Exclusion Criteria:

* Prior radiotherapy to the region of the study cancer within less than 6 months
* Patients who have received prior radiation therapy and who, in the opinion of the treating radiation oncologist, cannot be reirradiated safely without excess risk of severe toxicity given prior radiation dose to critical structures.
* Patients with known contraindications to radiotherapy, including inherited syndromes associated with hypersensitivity to ionizing radiation (e.g., Ataxia-Telangiectasia, Nijmegen Breakage Syndrome)
* Female patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-06-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction via qualitative interview and app based EMAs | 75 days
  Proportion of patients satisfied with the mHealth app. Patient satisfaction will be collected during the follow-up qualitative interview, and data will be analyzed using qualitative methods. The intervention will be deemed feasible if at least 75% of patients report that the app is easy to use and useful. Specifically, we will describe how often the app is used to measure symptoms, treatment effects, medication adherence, and pain, as well as HR-QOL and barriers to care.
Patient perceptions of mHealth platform | 75 days
  Proportion of patients who deem the mHealth app easy to use and useful. To gauge patient perception of mHealth platform with feedback from qualitative interview and app based EMAs. The final survey asks questions on the patients' thoughts, feelings, and opinions about the intervention they received over the course of the study.

SECONDARY OUTCOMES:
Feasibility of intervention | 75 days
  Proportion of patients who complete the phone-based surveys. Feasibility of the study will be determined by the proportion of participants who complete >/=75% of phone-based assessments. The app allows for the completion rate to be quantified.
Patient-reported barriers to care | 75 days
  Proportion of patients who report barriers to care as indicated by feedback from qualitative interview and app based EMAs.
Changes in weekly FACT-HN, FACT-Cx, or FACT-En scores over time | 75 days
  Proportion of changes in weekly FACT-HN, FACT-Cx, or FACT-En scores over time as indicated by feedback from qualitative interview and app based EMAs.
Completion rates of daily questionnaires | 75 days
  Proportion of daily questionnaires completed as indicated by EMA completion rate.

IPD SHARING:
Plan to Share IPD: No